CLINICAL TRIAL: NCT03717831
Title: Muscle Dysfunction and Functional Outcomes in Patients With and Surviving Critical Illness
Brief Title: Muscle Dysfunction in Critical Illness
Status: Completed | Type: Observational
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, Kirby Mayer, Graduate Research Assistant, University of Kentucky
Other Study IDs: 46072-58919
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Critical Illness; Intensive Care (ICU) Myopathy; PICS; Muscle Weakness
Keywords: muscle ultrasound; post-intensive care syndrome; physical function; muscle tissue analysis
MeSH Terms: conditions — Critical Illness; Muscular Diseases; Muscle Weakness; postintensive care syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy: Healthy subjects will be enrolled as age and activity matched controls for muscle power assessment at one time-point to establish normative values.
  Interventions: Other: Observational study of standard of care
- ICU: Observational, subjects enrolled initially in the ICU and followed for six months after hospital discharge. ICU subdivided based on diagnosis
  Interventions: Other: Observational study of standard of care

INTERVENTIONS:
Other: Observational study of standard of care — Observational cohort study

SUMMARY:
Patients surviving critical illness suffered significant skeletal muscle dysfunction and weakness that impacts their functionality and independence. The primary purpose of this project is to develop a classification system based on the health and function of the muscle at very early time points during critical illness. The investigators will determine if muscle ultrasound can predict functional recovery at six-months post hospital discharge. Researchers will assess muscle health and function from starting day one of admission to ICU and continue until six months of recovery. In addition to muscle ultrasound, the investigators will assess muscle strength and power, and perform muscle tissue analysis on a subset of individuals. These findings will be correlated to physical function and independence at six-month follow-up.

DETAILED DESCRIPTION:
Patients surviving critical illness experience significant skeletal muscle dysfunction and weakness. Muscle atrophy suffered during critical illness has a long-term impact on the functionality and mobility of these individuals.1-6 The underlying etiology is multifactorial, but largely thought to be caused by immobility(bed-rest), severity of illness, prolonged mechanical ventilation, sepsis, systematic inflammation, and delirium.7-9 Additionally, these alterations are purported to impair recovery of muscle function following discharge from the intensive care unit (ICU) leading to long-term physical deficits. From previous randomized controlled trials, results have demonstrated that early rehabilitation focused on mobility may positively influence patient functional outcomes.10 However, a number of randomized controlled trials implementing early rehabilitation fail to demonstrate robust immediate or long-term benefits.11,12 Mixed results may in large part be due to inconsistency in early assessment and classification of these patients.

In recent years, researchers have utilized ultrasound to classify and track changes in muscle size and quality; demonstrating up to 30% decline in rectus femoris cross-sectional area in the first ten days of critical illness.13,14 In addition, muscle tissue analysis have elucidated morphological changes including myofiber necrosis in 40% of patients with acute respiratory distress syndrome. In the recovery phase, tissue analysis revealed a reduction in satellite cells within the muscle, sparking the hypothesis that these individuals have an impaired regenerative capacity.15 The absence of satellite cells may not be responsible for alterations in recovery solely, if at all.16 The investigators propose that increased collagen production within the muscle tissue is a major contributor to impaired or slow recovery of muscle tissue. The investigators hypothesize that distinct phenotypes of patients exist with different activation of physiologic pathways and therefore different clinical and functional presentations. The primary purpose of this study is to develop a model to classify patients based on markers of muscle function, clinical composition, and functional data. This classification is multifactorial which will enable improved prediction of the patient's recovery trajectory at very early time-points.

Moreover, studies elucidating the underlying muscle biology and physiologic mechanisms have yet to connect those changes to physical function and independence. Correlating specific markers of muscle health to functional outcome measures is a necessary step to provide clinicians with evidence to support and adapt their practice in relation to the pathophysiology of the muscle. Finally, muscular power has not been examined in this population. Muscular power is a key component of functional mobility that is not a current focus in critical care rehabilitation. Power may be a primary culprit of reductions in functionality specifically related to performing simple task such as sit-to-stand with adequate strength and velocity. Studying power in this population is novel and could lead to immediate changes in rehabilitation practice.

Aim 1: Examine and quantify changes in muscular power during critical illness and through the first six months of recovery. Hypothesis: Patients with longer times immobilized and higher severity of illness will have larger declines in muscle power during hospitalization with slower recovery of muscle power in the first six months after discharge. To test this hypothesis, the investigators will longitudinally record muscular power using a linear transducer with a standardized weight-apparatus. This is an innovative approach and novel in this population.

Aim 2: Determine the relationship of the physical function and independence to muscle function. The correlation between characteristics of muscle health to patient's functional status has not been performed to this extent. Hypothesis: Patients with the steepest declines in rectus femoris muscle cross-sectional area in the first seven days of ICU admission will have lower scores of functional outcomes requiring higher levels of assistance at hospital discharge. Researchers will compare findings from muscle ultrasound (size and structure), muscle strength, muscle power, and functional endurance to functional outcomes during critical illness and across the first six months of recovery. These data will be analyzed and stratified based on predictive functional recovery trajectories.

Aim 3: Elucidate the molecular and cellular mechanisms leading to muscle dysfunction and impaired recovery following critical illness. Specifically, to determine the effect of myofiber type on functional capacity and explore the role of collagen and lipid deposition in the capacity for muscle to regenerate. Hypothesis: Patients with higher severity of illness that require more days on mechanical ventilation (MV) will have increased collagen production in the extra-cellular matrix leading to larger disability at 6-month follow-up. To test this hypothesis, muscular biopsies will be performed within two weeks of hospital discharge and again at 6 months post hospitalization.

This study builds the understanding that clinicians have the knowledge and resources to predict which patients will suffer the largest deficits. Thus, these classifications will enable clinicians to identify, at very early-timepoints, which patients will benefit from rehabilitation interventions. Furthermore, this proposal starts to address classifying patients based on phenotypes, including the concept of responders and non-responders. Establishing a multi-factorial classification system with components of muscle function will support rehabilitation clinicians in their decision to allocate early interventions. Streamlined allocation of interventions will mitigate the negative consequences of critical illness and maximize long-term patient outcomes

ELIGIBILITY:
Inclusion Criteria:

* admitted to medicine, cardio-thoracic or trauma ICU
* initial primary or secondary diagnosis of acute respiratory distress/failure
* mechanical ventilation (predicted for at-least 72 hours)

Exclusion Criteria:

* receiving palliative treatment
* attending physician excluding due to high-risk of mortality
* neurological injury or event
* lower extremity amputee
* pregnant
* non-ambulatory prior to admission

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to ICU for critical illness with diagnosis of acute respiratory failure will be enrolled in this observational study.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Physical function | 6 month follow-up
  Gait speed measured with 4 meter (Short Performance Physical Battery)

SECONDARY OUTCOMES:
Capacity for physical activity/exercise | 6 month follow-up
  Distance walked during 6 minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Kirby Mayer, DPT, PhD(c), Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bienvenu OJ, Colantuoni E, Mendez-Tellez PA, Dinglas VD, Shanholtz C, Husain N, Dennison CR, Herridge MS, Pronovost PJ, Needham DM. Depressive symptoms and impaired physical function after acute lung injury: a 2-year longitudinal study. Am J Respir Crit Care Med. 2012 Mar 1;185(5):517-24. doi: 10.1164/rccm.201103-0503OC. Epub 2011 Dec 8. PMID 22161158
- [Result] Fan E, Dowdy DW, Colantuoni E, Mendez-Tellez PA, Sevransky JE, Shanholtz C, Himmelfarb CR, Desai SV, Ciesla N, Herridge MS, Pronovost PJ, Needham DM. Physical complications in acute lung injury survivors: a two-year longitudinal prospective study. Crit Care Med. 2014 Apr;42(4):849-59. doi: 10.1097/CCM.0000000000000040. PMID 24247473
- [Result] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Result] Yang T, Li Z, Jiang L, Wang Y, Xi X. Risk factors for intensive care unit-acquired weakness: A systematic review and meta-analysis. Acta Neurol Scand. 2018 Aug;138(2):104-114. doi: 10.1111/ane.12964. Epub 2018 May 29. PMID 29845614
- [Result] Rawal G, Yadav S, Kumar R. Post-intensive Care Syndrome: an Overview. J Transl Int Med. 2017 Jun 30;5(2):90-92. doi: 10.1515/jtim-2016-0016. eCollection 2017 Jun. PMID 28721340
- [Result] Schweickert WD, Pohlman MC, Pohlman AS, Nigos C, Pawlik AJ, Esbrook CL, Spears L, Miller M, Franczyk M, Deprizio D, Schmidt GA, Bowman A, Barr R, McCallister KE, Hall JB, Kress JP. Early physical and occupational therapy in mechanically ventilated, critically ill patients: a randomised controlled trial. Lancet. 2009 May 30;373(9678):1874-82. doi: 10.1016/S0140-6736(09)60658-9. Epub 2009 May 14. PMID 19446324
- [Result] Morris PE, Berry MJ, Files DC, Thompson JC, Hauser J, Flores L, Dhar S, Chmelo E, Lovato J, Case LD, Bakhru RN, Sarwal A, Parry SM, Campbell P, Mote A, Winkelman C, Hite RD, Nicklas B, Chatterjee A, Young MP. Standardized Rehabilitation and Hospital Length of Stay Among Patients With Acute Respiratory Failure: A Randomized Clinical Trial. JAMA. 2016 Jun 28;315(24):2694-702. doi: 10.1001/jama.2016.7201. PMID 27367766
- [Result] Puthucheary ZA, Phadke R, Rawal J, McPhail MJ, Sidhu PS, Rowlerson A, Moxham J, Harridge S, Hart N, Montgomery HE. Qualitative Ultrasound in Acute Critical Illness Muscle Wasting. Crit Care Med. 2015 Aug;43(8):1603-11. doi: 10.1097/CCM.0000000000001016. PMID 25882765
- [Result] Dos Santos C, Hussain SN, Mathur S, Picard M, Herridge M, Correa J, Bain A, Guo Y, Advani A, Advani SL, Tomlinson G, Katzberg H, Streutker CJ, Cameron JI, Schols A, Gosker HR, Batt J; MEND ICU Group; RECOVER Program Investigators; Canadian Critical Care Translational Biology Group. Mechanisms of Chronic Muscle Wasting and Dysfunction after an Intensive Care Unit Stay. A Pilot Study. Am J Respir Crit Care Med. 2016 Oct 1;194(7):821-830. doi: 10.1164/rccm.201512-2344OC. PMID 27058306